CLINICAL TRIAL: NCT02679729
Title: A Phase I, Randomized, Single-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD5634 Following Single-Ascending Inhaled Doses (Part A) and After Single Inhaled and Intravenous Doses (Part B) in Healthy Subjects
Brief Title: To Assess the Safety, Tolerability and Pharmacokinetics of AZD5634 Following Inhaled and Intravenous (IV)Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D6600C00001
Record Dates: First submitted 2016-02-03; First posted 2016-02-10 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis
Keywords: inhaled dose; intravenous dose; healthy subjects; safety; tolerability; pharmacokinetics; AZD5634; jet nebulizer
MeSH Terms: conditions — Cystic Fibrosis | interventions — Inhalation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Part A, Dose Level 1 (Experimental): Subjects will inhale single doses of AZD5634 or placebo under fasted conditions and will rinse his/her mouth with approximately 100 mL (up to 240 mL) of water which must be swallowed
  Interventions: Drug: AZD5634 for inhalation; Other: Placebo
- Part A, Dose Level 2 (Experimental): Subjects will inhale single doses of AZD5634 or placebo under fasted conditions and will rinse his/her mouth with approximately 100 mL (up to 240 mL) of water which must be swallowed
  Interventions: Drug: AZD5634 for inhalation; Other: Placebo
- Part A, Dose Level 3 (Experimental): Subjects will inhale single doses of AZD5634 or placebo under fasted conditions and will rinse his/her mouth with approximately 100 mL (up to 240 mL) of water which must be swallowed
  Interventions: Drug: AZD5634 for inhalation; Other: Placebo
- Part A, Dose Level 4 (Experimental): Subjects will inhale single doses of AZD5634 or placebo under fasted conditions and will rinse his/her mouth with approximately 100 mL (up to 240 mL) of water which must be swallowed
  Interventions: Drug: AZD5634 for inhalation; Other: Placebo
- Part A, Dose Level 5 (Experimental): Subjects will inhale single doses of AZD5634 or placebo under fasted conditions and will rinse his/her mouth with approximately 100 mL (up to 240 mL) of water which must be swallowed
  Interventions: Drug: AZD5634 for inhalation; Other: Placebo
- Part A, Dose Level 6 (Experimental): Subjects will inhale single doses of AZD5634 or placebo under fasted conditions and will rinse his/her mouth with approximately 100 mL (up to 240 mL) of water which must be swallowed
  Interventions: Drug: AZD5634 for inhalation; Other: Placebo
- Part A, Dose Level 7 (Experimental): Subjects will inhale single doses of AZD5634 or placebo under fasted conditions and will rinse his/her mouth with approximately 100 mL (up to 240 mL) of water which must be swallowed
  Interventions: Drug: AZD5634 for inhalation; Other: Placebo
- Part B, Dose Level 1 (Experimental): Subjects will receive a single dose of IV AZD5634 and after a washout period of 14 days the same subjects will receive a single dose of inhaled AZD5634
  Interventions: Drug: AZD5634 for infusion

INTERVENTIONS:
Drug: AZD5634 for inhalation — Solution, citrate buffer, saline nebulizer solution; strength 0.1 - 5 mg/g; administered by jet nebulizer
  Arms: Part A, Dose Level 1; Part A, Dose Level 2; Part A, Dose Level 3; Part A, Dose Level 4; Part A, Dose Level 5; Part A, Dose Level 6; Part A, Dose Level 7
Drug: AZD5634 for infusion — Solution, citrate buffer, saline solution for infusion; strength 0.013 mg/mL
  Arms: Part B, Dose Level 1
Other: Placebo — inactive substance
  Arms: Part A, Dose Level 1; Part A, Dose Level 2; Part A, Dose Level 3; Part A, Dose Level 4; Part A, Dose Level 5; Part A, Dose Level 6; Part A, Dose Level 7

SUMMARY:
This is a Phase 1, first-in-human (FIH) single ascending dose study being conducted to better understand the safety, tolerability and pharmacokinetics of AZD5634 in healthy subjects

DETAILED DESCRIPTION:
This study is a Phase I, FIH, randomized, single-blinded (study center staff remain blinded during the dosing phase of the study), placebo-controlled, single ascending dose, sequential dose group study in healthy male subjects and/or female subjects of non-childbearing potential at a single study center to assess AZD5634 following inhaled and intravenous dose administration

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and/or female subjects aged 18 - 50 years with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at screening and on admission to the unit, must not be lactating and must be of non-childbearing potential, confirmed at screening by fulfilling 1 of the following criteria:

   * Post-menopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and follicle-stimulating hormone (FSH) levels in the post-menopausal range.
   * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but not tubal ligation.
4. Have a body mass index (BMI) between 18 and 30 kg/m2, inclusive, and weigh at least 50 kg and no more than 100 kg, inclusive.
5. Have a FEV1 (Forced expiratory volume in 1 second in liters) ≥ 80% of the predicted value at screening.
6. Provision of signed, written and dated informed consent for optional genetic/biomarker research.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the administration of investigational medicinal product (IMP).
4. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the investigator.
5. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV).
6. Abnormal vital signs, after 10 minutes supine rest, at screening and check-in, defined as any of the following:

   * Systolic blood pressure (SBP) < 90mmHg (millimeter of mercury) or ≥ 140 mmHg
   * Diastolic blood pressure (DBP) < 50mmHg or ≥ 90 mmHg
   * Heart Rate < 45 or > 85 beats per minute (bpm)
7. Any clinically significant abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically significant abnormalities in the 12-lead ECG, as considered by the investigator that may interfere with the interpretation of QTc (QT [ECG interval measured from the onset of the QRS complex to the end of the T wave] interval corrected for heart rate) interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy, at screening.
8. PR (PQ [ECG interval measured from the onset of the P wave to the onset of the QRS complex]) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation, at screening.
9. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS (ECG interval measured from the onset of the QRS complex to the J point) > 110 ms but < 115 ms are acceptable if there is no evidence of, for example, ventricular hypertrophy or pre-excitation, at screening.
10. Serum/plasma potassium levels are outside the normal range and lower than 3.5 to 5.1 mEq/L (milliequivalents per liter) at screening and prior to dosing.
11. Has active lung disease/asthma that requires treatment.
12. Known or suspected history of drug abuse, as judged by the investigator.
13. Current smokers or those who have smoked or used nicotine products within the previous 3 months.
14. History of alcohol abuse or excessive intake of alcohol, as judged by the investigator.
15. Positive screen for drugs of abuse, cotinine (nicotine), or alcohol at screening or admission to the unit.
16. History of severe allergy/hypersensitivity or ongoing clinically significant allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5634.
17. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea, chocolate), as judged by the investigator.
18. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the administration of IMP.
19. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the administration of IMP or longer if the medication has a long half-life.
20. Plasma donation within 1 month of screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening.
21. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the administration of IMP in this study. The period of exclusion is 3 months after the final dose from a previous study.

    Note: Subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.
22. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
23. Involvement of any Astra Zeneca, PAREXEL or study site employee or their close relatives.
24. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
25. Subjects who are vegans or have medical dietary restrictions.
26. Subjects who cannot communicate reliably with the investigator.

    In addition, any of the following is regarded as a criterion for exclusion from the genetic research:
27. Previous bone marrow transplant.
28. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MDCM, M.Sc, CPI, Principal Investigator — PAREXEL Early Phase Clinical Unit Baltimore
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Baltimore, Maryland

REFERENCES:
- [Derived] Kristensson C, Astrand A, Donaldson S, Goldwater R, Abdulai R, Patel N, Gardiner P, Tehler U, Mercier AK, Olsson M, Ersdal E, Maenpaa J, Bramer T, Malmgren A, Bennett W, Keen C. AZD5634, an inhaled ENaC inhibitor, in healthy subjects and patients with cystic fibrosis. J Cyst Fibros. 2022 Jul;21(4):684-690. doi: 10.1016/j.jcf.2022.02.010. Epub 2022 Feb 26. PMID 35227647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 1, first-in-human (FIH), single-blind, placebo-controlled, single ascending dose (SAD), sequential dose group study in healthy male participants and female participants of non-childbearing potential at 2 study centers (EPCU Baltimore and EPCU Los Angeles). The study comprised of Part A and Part B.
Pre-assignment Details: The study consisted of a screening period (Days -28 to -1).
Groups:
- Part A - AZD5634 - 10 μg: Participants received inhaled single doses of AZD5634 10 μg under fasted conditions
- Part A - AZD5634 27 μg: Participants received inhaled single doses of AZD5634 27 μg under fasted conditions
- Part A - AZD5634 81 μg: Participants received inhaled single doses of AZD5634 81 μg under fasted conditions
- Part A - AZD5634 216 μg: Participants received inhaled single doses of AZD5634 216 μg under fasted conditions
- Part A - AZD5634 648 μg: Participants received inhaled single doses of AZD5634 648 μg under fasted conditions
- Part A - AZD5634 1296 μg: Participants received inhaled single doses of AZD5634 1296 μg under fasted conditions
- Part A - AZD5634 1692 μg: Participants received inhaled single doses of AZD5634 1692 μg under fasted conditions
- Part A - Placebo: 2 participants per dose level received single dose of placebo in Part A
- PartB- AZD5634-Intravenous(IV) 65μg and Inhalation(IN) 1692μg: After safety evaluation of all inhaled AZD5634 cohorts, 6 participants (who did not participate in Part A) were admitted for inhaled (1692 μg AZD5634) and IV (65 μg AZD5634) dosing (fixed dosing; IV first followed by inhalation), with at least a 14 day washout between dosing
Period: Overall Study
Arm/Group | Part A - AZD5634 - 10 μg | Part A - AZD5634 27 μg | Part A - AZD5634 81 μg | Part A - AZD5634 216 μg | Part A - AZD5634 648 μg | Part A - AZD5634 1296 μg | Part A - AZD5634 1692 μg | Part A - Placebo | PartB- AZD5634-Intravenous(IV) 65μg and Inhalation(IN) 1692μg
Started | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 14 | 6
Completed | 6 | 5 | 6 | 6 | 5 | 6 | 5 | 14 | 6
Not Completed | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant decision | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AZD5634 - Inhaled 10 μg: Participants received inhaled single doses of AZD5634 10 μg under fasted conditions
- AZD5634 27 μg: Participants received inhaled single doses of AZD5634 27 μg under fasted conditions
- AZD5634 81 μg: Participants received inhaled single doses of AZD5634 81 μg under fasted conditions
- AZD5634 216 μg: Participants received inhaled single doses of AZD5634 216 μg under fasted conditions
- AZD5634 648 μg: Participants received inhaled single doses of AZD5634 648 μg under fasted conditions
- AZD5634 1296 μg: Participants received inhaled single doses of AZD5634 1296 μg under fasted conditions
- AZD5634 1692 μg: Participants received inhaled single doses of AZD5634 1692 μg under fasted conditions
- Placebo: 2 participants per dose level received single dose of placebo in Part A
- AZD5634 - IV 65 μg and IN 1692 μg: After safety evaluation of all inhaled AZD5634 cohorts, 6 participants (who did not participate in Part A) were admitted for inhaled (1692 μg AZD5634) and IV (65 μg AZD5634) dosing (fixed dosing; IV first followed by inhalation), with at least a 14 day washout between dosing
- Total: Total of all reporting groups
Arm/Group | AZD5634 - Inhaled 10 μg | AZD5634 27 μg | AZD5634 81 μg | AZD5634 216 μg | AZD5634 648 μg | AZD5634 1296 μg | AZD5634 1692 μg | Placebo | AZD5634 - IV 65 μg and IN 1692 μg | Total
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 14 | 6 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Data for Part A and Part B are presented in separate rows. Part A and Part B data when added (57 + 6) will give the overall total of 63
  Years
    Part A: number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 14 | 0 | 57
    Part A | 36.5 (12.2) | 33.3 (9.3) | 31.8 (3.4) | 32.0 (6.9) | 37.7 (9.1) | 31.7 (5.2) | 35.2 (10.6) | 32.6 (8.9) |  | 34.0 (8.3)
    Part B: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
    Part B |  |  |  |  |  |  |  |  | 32.0 (7.9) | 32.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3
  Male | 6 | 7 | 6 | 6 | 5 | 6 | 5 | 13 | 6 | 60

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of AZD5634 Following Inhaled Administration of Single-ascending Doses (SAD) (Part A) and Following Administration of Single Inhaled and IV Doses (Part B).
Description: To assess the safety and tolerability of AZD5634 in terms of number of participants following inhaled administration of single-ascending doses (SAD) (Part A) and following administration of single inhaled and IV doses (Part B)
Time Frame: Screening (serious adverse event, SAE), Day -1 (SAE), Spontaneous plus Predose, 3,12,24, and 48 h postdose (Days 1 to 3), Follow-up 7-10 days postdose, 2 months post final dose.
Population: All partcipants in safety analysis set who received at least 1 dose of IMP and for whom any safety post-dose data were available were included in the safety analysis for the study.
Measure: Number; unit: Participants
Groups:
- Part A - AZD5634 10 µg: Participants received inhaled single doses of AZD5634 10 µg under fasted conditions
- Part A - AZD5634 27 µg: Participants received inhaled single doses of AZD5634 27 µg under fasted conditions
- Part A - AZD5634 81 µg: Participants received inhaled single doses of AZD5634 81 µg under fasted conditions
- Part A - AZD5634 216 µg: Participants received inhaled single doses of AZD5634 216 µg under fasted conditions
- Part A - AZD5634 648 µg: Participants received inhaled single doses of AZD5634 648 µg under fasted conditions
- Part A - AZD5634 1296 µg: Participants received inhaled single doses of AZD5634 1296 µg under fasted conditions
- Part A - AZD5634 1692 µg: Participants received inhaled single doses of AZD5634 1692 µg under fasted conditions
- Part A - Placebo for AZD5634: 2 participants per dose level received single dose of placebo in Part A
- Part B - AZD5634 IV 65 µg: Participants received IV dose of AZD5634 65 µg
- Part B - AZD5634 IN 1692 µg: Participants received an IV dose and after a washout period of 14 days this was followed by an inhaled dose AZD5634 1692 µg to the same participants
Arm/Group | Part A - AZD5634 10 µg | Part A - AZD5634 27 µg | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part A - Placebo for AZD5634 | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 6 | 6 | 6 | 14 | 6 | 6
Participants
  Any AE during treatment | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 3 | 2 | 1
  Any AE with outcome = death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE (including events with outcome = death) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AE during Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Observed Maximum Plasma Concentration, Taken Directly From the Individual Concentration-time Curve (Cmax)- For Part A and Part B
Description: To assess the pharmacokinetic (PK) parameter Cmax of AZD5634 following single-dose inhalation administration of AZD5634 in Part A and following single-dose IV or inhalation administration of AZD5634 in Part B. Note: Due to the participant and/or data exclusion described above, there are no PK data available for the 10 μg dose cohort and very limited data for the 27 μg dose cohort. Therefore, these 2 cohorts were not included in PK results interpretation and summary statistics.
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: The PK analysis set for Part A consisted of participants in the safety analysis set who received AZD5634 and for Part B consisted of participants who completed both treatment periods and for whom at least one of the PK parameters Cmax, AUC0-t or AUC were calculated, with no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 6 | 6
nmol/L | 0.01605 (18.8) | 0.04581 (45.2) | 0.2977 (20.0) | 0.3043 (46.5) | 0.5316 (51.6) | 6.070 (8.9) | 0.3808 (34.7)
Statistical Analysis 1: Comparison: Part A - AZD5634 81 µg vs Part A - AZD5634 216 µg vs Part A - AZD5634 648 µg vs Part A - AZD5634 1296 µg vs Part A - AZD5634 1692 µg; Statistical Analysis for Part A; Test type: Superiority or Other; Slope = 0.625, 95% CI 2-sided [0.396 to 0.853]

3. Secondary Outcome: Area Under Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC) for Part A and Part B
Description: To assess the pharmacokinetic parameter AUC of AZD5634 following single-dose inhalation administration of AZD5634 in Part A and following single-dose IV or inhalation administration of AZD5634 in Part B. AUC was estimated by AUC(0-last) + Clast/λz where Clast was the last observed quantifiable concentration. AUCs were calculated using the linear trapezoidal method when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing. AUC0-t is expanded as area under the plasma concentration-time curve from time zero to time of last quantifiable concentration. Note:Due to the participant and/or data exclusion described above, there are no PK data available for the 10 μg dose cohort and very limited data for the 27 μg dose cohort. Therefore, these 2 cohorts were not included in PK results interpretation and summary statistics.
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 6 | 6
h*nmol/L | NA (NA) — Due to the participant and/or data exclusion, data were not available | 0.1757 (34.9) | 1.258 (16.7) | 1.299 (57.2) | 2.837 (71.5) | 2.329 (11.3) | 1.777 (37.2)
Statistical Analysis 1: Comparison: Part A - AZD5634 81 µg vs Part A - AZD5634 216 µg vs Part A - AZD5634 648 µg vs Part A - AZD5634 1296 µg vs Part A - AZD5634 1692 µg; Statistical Analysis for Part A; Test type: Superiority or Other; Slope = 1.20, 95% CI 2-sided [0.905 to 1.49]

4. Secondary Outcome: Area Under the Plasma Concentration-curve From Time Zero to Time of Last Quantifiable Concentration [AUC(0-t)] for Part A and Part B
Description: To assess the pharmacokinetic parameter AUC(0-t) of AZD5634 following single-dose inhalation administration of AZD5634 in Part A and following single-dose IV or inhalation administration of AZD5634 in Part B. Note: Due to the participant and/or data exclusion described above, there are no PK data available for the 10 μg dose cohort and very limited data for the 27 μg dose cohort. Therefore, these 2 cohorts were not included in PK results interpretation and summary statistics.
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 6 | 6
h*nmol/L | 0.01920 (60.1) | 0.1120 (62.2) | 1.301 (22.0) | 1.244 (57.2) | 2.664 (60.9) | 2.318 (11.4) | 1.831 (38.0)
Statistical Analysis 1: Comparison: Part A - AZD5634 81 µg vs Part A - AZD5634 216 µg vs Part A - AZD5634 648 µg vs Part A - AZD5634 1296 µg vs Part A - AZD5634 1692 µg; Statistical Analysis for Part A; Test type: Superiority or Other; Slope = 1.55, 95% CI 2-sided [1.34 to 1.76]

5. Secondary Outcome: Absolute Systemic Bioavailability After Inhalation (Part B Only) (Finhalation,Total)
Description: To assess the Absolute systemic bioavailability after inhalation (%), calculated separately as 100*AUCinhalation*Doseiv/(AUCiv*Doseinhalation)
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: The PK analysis set for Part B consisted of all participants who completed both treatment periods and for whom at least one of the PK parameters Cmax, AUC0-t or AUC were calculated in each treatment period, with no major protocol deviations thought to impact on the analysis of the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of bioavailable dose
Arm/Group | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 6 | 6
Percentage of bioavailable dose | NA (NA) — Due to the participant and/or data exclusion, data were not available | 2.928 (42.2)

6. Secondary Outcome: Renal Clearance (CLR), Estimated by Dividing Ae(0-last) by AUC0-t - For Part A and Part B
Description: To assess the pharmacokinetic parameter CLR of AZD5634 following single-dose inhalation administration of AZD5634 in Part A and following single-dose IV or inhalation administration of AZD5634 in Part B. Note: Due to the participant and/or data exclusion described above, there are no PK data available for the 10 μg dose cohort and very limited data for the 27 μg dose cohort. Therefore, these 2 cohorts were not included in PK results interpretation and summary statistics.
Time Frame: -12-0, 0-6, 6-12, 12-24, 24-48 h (Days 1 to 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 6 | 6
L/h | 1.449 (0.1332) | 0.8099 (0.2849) | 0.5828 (0.1724) | 0.9063 (0.2459) | 0.7333 (0.1893) | 0.6247 (0.3373) | 0.6939 (0.1044)

7. Secondary Outcome: Cmax, Divided by the Dose Aministered (Cmax/Dose) - For Part A and Part B
Description: To assess the pharmacokinetic parameter Cmax/Dose of AZD5634 following single-dose inhalation administration of AZD5634 in Part A and following single-dose IV or inhalation administration of AZD5634 in Part B. Note: Due to the participant and/or data exclusion described above, there are no PK data available for the 10 μg dose cohort and very limited data for the 27 μg dose cohort. Therefore, these 2 cohorts were not included in PK results interpretation and summary statistics.
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L/umol
Arm/Group | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 6 | 6
nmol/L/umol | 0.1473 (18.8) | 0.1576 (45.2) | 0.3415 (20.0) | 0.1745 (46.5) | 0.2335 (51.6) | 69.41 (8.9) | 0.1673 (34.7)

8. Secondary Outcome: Terminal Half-life (t1/2λz), Estimated as (ln2)/λz - For Part A and Part B
Description: To assess the pharmacokinetic parameter t1/2λz of AZD5634 following single-dose inhalation administration of AZD5634 in Part A and following single-dose IV or inhalation administration of AZD5634 in Part B. Note: Due to the participant and/or data exclusion described above, there are no PK data available for the 10 μg dose cohort and very limited data for the 27 μg dose cohort. Therefore, these 2 cohorts were not included in PK results interpretation and summary statistics.
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 6 | 6
Hours | NA (NA) — Due to the participant and/or data exclusion, data were not available | 1.519 (0.1499) | 1.903 (0.4722) | 3.144 (2.250) | 7.552 (5.438) | 0.1923 (0.05567) | 3.184 (1.816)

9. Secondary Outcome: AUC0-t, Divided by the Dose Administered (AUC0-t/Dose) - For Part A and Part B
Description: To assess the pharmacokinetic parameter AUC0-t/Dose of AZD5634 following single-dose inhalation administration of AZD5634 in Part A and following single-dose IV or inhalation administration of AZD5634 in Part B. Note: Due to the participant and/or data exclusion described above, there are no PK data available for the 10 μg dose cohort and very limited data for the 27 μg dose cohort. Therefore, these 2 cohorts were not included in PK results interpretation and summary statistics.
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L/umol
Arm/Group | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 6 | 6
h*nmol/L/umol | 0.1762 (60.1) | 0.3856 (62.2) | 1.492 (22.0) | 0.7137 (57.2) | 1.170 (60.9) | 26.51 (11.4) | 0.8044 (38.0)

10. Secondary Outcome: AUC, Divided by the Dose Administered (AUC/Dose) - For Part A and Part B
Description: To assess the pharmacokinetic parameter AUC/Dose of AZD5634 following single-dose inhalation administration of AZD5634 in Part A and following single-dose IV or inhalation administration of AZD5634 in Part B. Note: Due to the participant and/or data exclusion described above, there are no PK data available for the 10 μg dose cohort and very limited data for the 27 μg dose cohort. Therefore, these 2 cohorts were not included in PK results interpretation and summary statistics.
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L/umol
Arm/Group | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 6 | 6
h*nmol/L/umol | NA (NA) — Due to the participant and/or data exclusion, data were not available | 0.6046 (34.9) | 1.444 (16.7) | 0.7450 (57.2) | 1.246 (71.5) | 26.63 (11.3) | 0.7805 (37.2)

11. Secondary Outcome: Systemic Clearance for AZD5634 Estimated as Dose Divided by AUC (Part B IV Dosing Only) (CL)
Description: To assess the pharmacokinetic parameter CL of AZD5634 following single-dose IV administration of AZD5634 in Part B
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part B - AZD5634 IV 65 µg
Number analyzed (Participants) | 6
L/h | 37.74 (4.220)

12. Secondary Outcome: Apparent Clearance for AZD5634 Estimated as Dose Divided by AUC (Part A and Part B Inhaled Dosing Only) (CL/F)
Description: To assess the pharmacokinetic parameter CL/F of AZD5634 following single-dose inhalation administration of AZD5634 in Part A and following single-dose inhalation administration of AZD5634 in Part B. Note: Due to the participant and/or data exclusion described above, there are no PK data available for the 10 μg dose cohort and very limited data for the 27 μg dose cohort. Therefore, these 2 cohorts were not included in PK results interpretation and summary statistics.
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 6
L/h | NA (NA) — Due to the participant and/or data exclusion, data were not available | 1727 (589.7) | 699.9 (115.3) | 1518 (852.7) | 929.8 (548.2) | 1346 (457.8)

13. Secondary Outcome: Mean Residence Time (MRT) - For Part A and Part B
Description: To assess the pharmacokinetic parameter MRT of AZD5634 following single-dose inhalation administration of AZD5634 in Part A and following single-dose IV or inhalation administration of AZD5634 in Part B. Note: Due to the participant and/or data exclusion described above, there are no PK data available for the 10 μg dose cohort and very limited data for the 27 μg dose cohort. Therefore, these 2 cohorts were not included in PK results interpretation and summary statistics.
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 6 | 6
hour | NA (NA) — Due to the participant and/or data exclusion, data were not available | 2.742 (0.1741) | 3.529 (0.5093) | 4.157 (1.166) | 6.000 (2.009) | 0.1928 (0.02455) | 4.428 (1.293)

14. Secondary Outcome: Mean Absorption Time, Calculated as MRTinhaled - MRTIV (Part B Only) (MAT)
Description: To assess the pharmacokinetic parameter MAT of AZD5634 following single-dose IV or inhalation administration of AZD5634 in Part B
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 6 | 6
hour | NA (NA) — This parameter analysis was not applicable for this arm. | 4.236 (1.302)

15. Secondary Outcome: Volume of Distribution for AZD5634 at Steady State (IV Administration), Estimated by Dividing the MRT by the Systemic CL (Part B IV Dosing Only) (Vss)
Description: To assess the pharmacokinetic parameter Vss of AZD5634 following single-dose IV administration of AZD5634 in Part B
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Part B - AZD5634 IV 65 µg
Number analyzed (Participants) | 6
Litre | 7.202 (0.3915)

16. Secondary Outcome: Volume of Distribution for AZD5634 at Terminal Phase (IV Administration), Estimated by Dividing the Systemic CL by λz (Part B IV Dosing Only) (Vz)
Description: To assess the pharmacokinetic parameter Vz of AZD5634 following single-dose IV administration of AZD5634 in Part B
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Part B - AZD5634 IV 65 µg
Number analyzed (Participants) | 6
Litre | 10.25 (1.804)

17. Secondary Outcome: Apparent Volume of Distribution for AZD5634 at Terminal Phase (Inhaled Administration), Estimated by Dividing the CL/F by λz (Part A and Part B Inhaled Dosing Only) (Vz/F)
Description: To assess the pharmacokinetic parameter Vz/F of AZD5634 following single-dose inhalation administration of AZD5634 in Part A and Part B. Note: Due to the participant and/or data exclusion described above, there are no PK data available for the 10 μg dose cohort and very limited data for the 27 μg dose cohort. Therefore, these 2 cohorts were not included in PK results interpretation and summary statistics.
Time Frame: At predose, at 5, 15 and 30 min and at 1, 2, 3, 4, 6, 8, 12, 24, 36 and 48 h postdose (Days 1 to 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part B - AZD5634 IN 1692 µg
Number analyzed (Participants) | 3 | 5 | 5 | 6 | 5 | 6
Litre | NA (NA) — Due to the participant and/or data exclusion, data were not available | 3775 (1306) | 1864 (178.2) | 5416 (1905) | 7115 (2202) | 5361 (1077)

ADVERSE EVENTS:
Time Frame: Screening (SAE), Day -1 (SAE), Spontaneous plus Predose, 3,12,24, and 48 h postdose (Days 1 to 3), Follow-up 7-10 days postdose, 2 months post final dose.
Groups:
- Part B - AZD5634 IV 65 µg: Participants received IV dose of IV 65 µg
- Part B - AZD5634 IN 1692 µg: Participants received IV dose and after a washout period of 14 days this was followed by an inhaled dose AZD5634 1692 µg to the same participants
Arm/Group | Part A - AZD5634 10 µg | Part A - AZD5634 27 µg | Part A - AZD5634 81 µg | Part A - AZD5634 216 µg | Part A - AZD5634 648 µg | Part A - AZD5634 1296 µg | Part A - AZD5634 1692 µg | Part A - Placebo for AZD5634 | Part B - AZD5634 IV 65 µg | Part B - AZD5634 IN 1692 µg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/14 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/7 | 0/6 | 1/6 | 1/6 | 0/6 | 2/6 | 3/14 | 2/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - AZD5634 10 µg (N=6) | Part A - AZD5634 27 µg (N=7) | Part A - AZD5634 81 µg (N=6) | Part A - AZD5634 216 µg (N=6) | Part A - AZD5634 648 µg (N=6) | Part A - AZD5634 1296 µg (N=6) | Part A - AZD5634 1692 µg (N=6) | Part A - Placebo for AZD5634 (N=14) | Part B - AZD5634 IV 65 µg (N=6) | Part B - AZD5634 IN 1692 µg (N=6)
Medical device site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential and property of the sponsor. No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB.